CLINICAL TRIAL: NCT03502759
Title: Improving Patient Communication About SUDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Child Neurology Foundation (Unknown); Greenwich Biosciences (Industry)
Responsible Party: Principal Investigator, Randall Grout, MD, Faculty, Ped Health Services, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1803547954
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: SUDEP; Epilepsy
Keywords: SUDEP; Epilepsy
MeSH Terms: conditions — Sudden Unexpected Death in Epilepsy; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Seizure patients receive usual care.
- Post-intervention (Experimental): Physicians provide care enhanced by computer based clinical decision support about SUDEP.
  Interventions: Behavioral: CHICA SUDEP module

INTERVENTIONS:
Behavioral: CHICA SUDEP module — CHICA reminds physicians to counsel patients/families about the risk of SUDEP.
  Arms: Post-intervention

SUMMARY:
Children with generalized tonic-clonic seizures (GTCS) have about a 1 in 4500 of succumbing to sudden unexpected death in epilepsy (SUDEP). For that reason, the American Academy of Neurology recommends that clinicians caring for these children make their families aware of this small but important risk and provide appropriate supportive follow-up resources. Moreover, existing evidence suggests that children with poorly controlled GTCS have a strikingly increased odds of SUDEP, 3-24 fold, raising the importance of improving seizure control.

Clinicians caring for these patients have multiple issues to address in the typical visit. The investigators propose to use information technology to help providers assure that addressing SUDEP is incorporated into their routine care. The investigators have developed the Child Health Improvement through Computer Automation system (CHICA), a computer based clinical decision support system for pediatric care. CHICA captures patient reported data in the waiting room and prioritizes clinical advice to the physician through the electronic health record (EHR).

CHICA is used in five primary care clinics in the Eskenazi health system where it supports general pediatric care. The goal of this project is to test the effectiveness of a SUDEP module in this setting where CHICA is already in use - with a future goal of developing a full suite of CHICA modules for child neurologists.

DETAILED DESCRIPTION:
Specifically, the investigators propose the following:

Aim 1: Add a "SUDEP module" to CHICA to identify children at increased risk of SUDEP, provide patient education materials that the clinician can share with the families, and recommend timelier follow-up with a child neurologist. The SUDEP module will be added to the existing installation of CHICA in the Eskenazi Health System in Indianapolis, IN so that SUDEP risk screening and advice are generated automatically in the setting of routine primary care in the 5 Eskenazi clinics.

Aim 2: Interview families of patients with epilepsy to determine if their pediatricians shared the SUDEP information and/or referred them to their neurologist. Families whose children are at risk for SUDEP will be identified through CHICA. The investigators will utilize the Pediatric Practice-based Research Network (PResNet) to follow-up these families by phone after their visits with the pediatrician. PResNet will determine if SUDEP was discussed, if a handout was provided, and if SUDEP has been discussed previously by their pediatrician or neurologist.

Aim 3: The investigators will assess physician and staff satisfaction regarding the SUDEP module of CHICA. Each year, PResNet will conduct a satisfaction survey among the clinic physicians and staff that use CHICA. The survey consists of general questions about CHICA that are asked every year and module-specific questions about new functionality that has been added.

ELIGIBILITY:
Inclusion Criteria:

Parent or Guardian of a child seen at one of five clinics in the Eskenazi health care system for which the child has had at least 2 lifetime motor seizures.

Exclusion Criteria:

Inability of the subject to understand the survey

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Parent recall of SUDEP counseling | within 2 weeks of a clinical encounter
  Parents will be contacted by phone and answer survey questions about SUDEP counseling during their child's most recent pediatric visit.

SECONDARY OUTCOMES:
Knowledge and comfort in taking care of child's epilepsy | within 2 weeks of a clinical encounter
  Parents will be contacted by phone and answer survey questions about their knowledge and comfort in taking care of their child's epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Randall W Grout, MD, Principal Investigator — Indiana University - Ped Health Services
Locations (1):
- Indiana University - Children's Health Services Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grout RW, Buchhalter J, Patel AD, Brin A, Clark AA, Holmay M, Story TJ, Downs SM. Improving Patient-Centered Communication about Sudden Unexpected Death in Epilepsy through Computerized Clinical Decision Support. Appl Clin Inform. 2021 Jan;12(1):90-99. doi: 10.1055/s-0040-1722221. Epub 2021 Feb 17. PMID 33598905